CLINICAL TRIAL: NCT05810194
Title: Retrospective Cohort Study Comparing a Novel Silicone Gel Wound Dressing vs Standard of Care in the Treatment of Radiation Dermatitis
Brief Title: Retrospective Cohort Study Comparing a Novel Gel Dressing vs SoC in the Treatment of Radiation Dermatitis
Status: Completed | Type: Observational
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: SPASX020
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Petrolatum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- StrataXRT
  Interventions: Device: StrataXRT
- Standard of care
  Interventions: Drug: Calendula; Drug: Aquaphor

INTERVENTIONS:
Device: StrataXRT — StrataXRT® is a TGA-approved silicone-based topical preparation. StrataXRT is a self-drying, non-sticky, transparent, silicone gel formulation and when used as directed, dries to form an inert, thin, flexible wound dressing with a protective layer that is gas permeable and waterproof. It is the only self-drying topical silicone gel indicated for the use on radiation dermatitis, which hydrates and protects compromised skin areas and open wounds from chemical and microbial invasion. StrataXRT helps create an optimal wound healing environment which leads to faster re-epithelialization and a reduced inflammatory response. The product can be applied to fresh incisions and excisions, open wounds and compromised skin surfaces.
  Groups: StrataXRT
Drug: Calendula — Calendula creams are over-the-counter (OTC) skin care ointments that are non-greasy, non-sticky, and quickly absorbed by the skin. Calendula is a topical agent derived from a plant of the marigold family Calendula Officinalis and is used in cuts, scrapes, chafing and minor burns. Containing numerous polyphenolic antioxidants, calendula has been studied in both the laboratory and clinical setting for the use in treating and preventing radiation induced skin toxicity.
  Groups: Standard of care
Drug: Aquaphor — Aquaphor, containing 41 percent petrolatum (or petroleum jelly), temporarily protects minor cuts, scrapes, and burns; Aquaphor protects and helps relieve chapped or cracked skin and lips, as well as helps protecting from the drying effects of wind and cold weather.
  Groups: Standard of care

SUMMARY:
Routinely collected data on radiation-induced skin toxicity from 2010 to 2022 will be retrospectively analyzed. Data will be split into two cohorts: patients that received 1) StrataXRT and 2) standard of care. The incidence of grade ≥ 2 radiation dermatitis, the time to onset of grade ≥ 2 radiation dermatitis, the radiation dose at onset of grade ≥ 2 radiation dermatitis, the incidence of moist desquamation and the number of treatment interruptions will be compared between the cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Head and Neck cancer treated with radiation therapy with or without chemotherapy
* Fractionated courses including at least 30 fractions (treatments)
* Minimum of 18 completed radiation treatments
* Radiation dose: > 50 Gy
* Radiation technique: IMRT
* Radiation equipment: TrueBeam or Tomotherapy

Exclusion Criteria:

* Prior radiation to the treatment area
* Patients with any medical condition such as active connective tissue disorder that predisposes them to an increased risk of potentially severe radiation dermatitis.
* Patients undergoing SBRT
* Patients with existing rashes or wounds in the target region or radiation therapy at RT start
* Patients receiving hypofractionation
* Patient receiving bolus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer patients treated with radiation therapy at UCLA from 2010 to 2022
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
CTCAE for Radiation Dermatitis | 5 weeks
  Acute radiation dermatitis measured weekly during radiotherapy treatment, using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 score (grade 0 - 5). A higher grade is considered a worse outcome.

SECONDARY OUTCOMES:
CTCAE for Hyperpigmentation | 5 weeks
  Acute hyperpigmentation measured weekly during radiotherapy treatment, using the Common Terminology Criteria for Adverse Events (CTCAE) score (grade 0 - 2). A higher grade is considered a worse outcome.
Number of patients requiring burn cream application | 5 weeks
  Total number of patients that required burn cream application during radiotherapy
Interval between radiotherapy start and burn cream application | 5 weeks
  Number of days between initiation of radiation therapy and first application of burn cream during radiotherapy
Number of patients requiring Mepilex application | 5 weeks
  Total number of patients that required Mepilex application during radiotherapy
Interval between radiotherapy start and Mepilex application | 5 weeks
  Number of days between initiation of radiation therapy and first application of Mepilex during radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, California, United States